CLINICAL TRIAL: NCT00854282
Title: The Role of Regulatory T Cell in Ovarian Cancer: Focus on Relationship Between
Brief Title: The Role of Regulatory T Cell in Ovarian Cancer: Focus on Relationship Between Clinical Prognosis and Regulatory T Cell Expression
Acronym: Tregs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Wen-Fang Cheng/Associate Professor, National Taiwan Unviersity Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 200812139R
Record Dates: First submitted 2009-03-01; First posted 2009-03-03 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Staging surgery or debulking surgery — Staging surgery or debulking surgery

SUMMARY:
Cancer is the leading cause of mortality in our country, and ovarian cancer becomes a more and more important disease gradually in the field of gynecologic malignancies. According to the statistics of the Department of Health, the incidence of ovarian cancer increased in recent years and the mortality rate was the highest among all gynecologic malignancies in Taiwan. Early diagnosis for ovarian cancer is difficult due to the lack of obvious and specific initial symptoms. Therefore, it is usually at advanced stage when the diagnosis is confirmed. The prognostic parameters for ovarian cancer include tumor stage, histological subtype and grade, residual tumor after surgical intervention and the response to chemotherapy. However, the possible mechanism of ovarian cancer is still not clear now, which has considerable influence on the management and prognosis of the patients.

Malignancy is considered as a multi-factorial disease, and the influence of immunologic mechanism on progression and prognosis of cancer is more and more important. The natural CD25+CD4+ regulatory T cells actively suppress pathologic and physiological immune response, contributing to the maintenance of immunological self-tolerance and immune homeostasis. The development and function of regulatory T cells depend on the expression of the transcription factor forkhead box P3 (FOXP3). The mechanisms of suppression are still not known well. Whatever the mechanisms of suppression are, it is necessary to control the magnitude of regulatory T cells-mediated suppression for the benefit of the host because too much suppression might lead to immunosuppression and render the host susceptible to infection and cancer.

We will collect the tumor tissue, ascites and peripheral blood during operation. Through this research we will set up the immunological profiles in the changes of lymphocytes, humoral immunity and cell-mediated immunity in ovarian cancer patients. The kinetic changes and associations between regulatory T cells and the severity and progression of disease will also be evaluated. Therefore, the role of regulatory T cells would be defined in the patients with ovarian cancer. We will also correlate the regulatory T cells with the clinical prognosis of ovarian cancer patients. Finally, we will try to find an efficient therapeutic strategy for the cancer patients.

DETAILED DESCRIPTION:
Methods:

All of the patients received four to six courses of adjuvant platinum-containing chemotherapy.Histologic grading was according to International Union against Cancer criteria (28). The stage of disease was classified according to the International Federation of Gynecology and Obstetrics (FIGO, 1987). Pelvic and paraaortic lymph node samplings will be performed, if the disease will be confined to within the ovary or will be without a ruptured capsule. The histopathologic data, including histologic type and histologic grade, will be evaluated by a certified pathologist. The maximal diameter of the residual tumor after surgery will be also recorded. All patients will be followed up at 3-month intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ovarian carcinoma who undergo hysterectomy, bilateral oophorectomy and tubal resection, omentectomy, and appendectomy will be enrolled and the clinical data will be obtained from our hospital.

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-01 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | from disease diagnosis to death

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan